CLINICAL TRIAL: NCT03777657
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Clinical Study Comparing the Efficacy and Safety of Tislelizumab (BGB-A317) Plus Platinum and Fluoropyrimidine Versus Placebo Plus Platinum and Fluoropyrimidine as First-Line Treatment in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Tislelizumab in Combination With Chemotherapy as First-Line Treatment in Adults With Inoperable, Locally Advanced or Metastatic Gastric, or Gastroesophageal Junction Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BGB-A317-305; 2018-000312-24 (EudraCT Number); CTR20181841 (Registry Identifier: ChinaDrugTrials); JapicCTI-194799 (Registry Identifier: Japic)
Record Dates: First submitted 2018-11-09; First posted 2018-12-17 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Gastric, or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — tislelizumab; Cisplatin; Oxaliplatin; Capecitabine; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + Chemotherapy (Experimental): Participants received 200 mg of tislelizumab intravenously with investigator's choice of chemotherapy once every 3 weeks for up to six treatment cycles. Chemotherapy consisted of 1000 mg/m² capecitabine twice daily on Days 1-14 and 130 mg/m² oxaliplatin on Day 1, or 800 mg/m² 5-fluorouracil (5-FU) on Days 1-5 and 80 mg/m² cisplatin on Day 1 of each 21-day cycle. Thereafter, participants continued treatment with 200 mg tislelizumab, with optional maintenance capecitabine (only permitted for participants who initially received capecitabine and oxaliplatin) once every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Oxaliplatin; Drug: Capecitabine; Drug: 5-Fluorouracil
- Placebo + Chemotherapy (Placebo Comparator): Participants received placebo intravenously with investigator's choice of chemotherapy once every 3 weeks for up to six treatment cycles. Chemotherapy consisted of 1000 mg/m² capecitabine twice daily on Days 1-14 and 130 mg/m² oxaliplatin on Day 1, or 800 mg/m² 5-FU on Days 1-5 and 80 mg/m² cisplatin on Day 1 of each 21-day cycle. Thereafter, participants continued treatment with placebo with optional maintenance capecitabine (only permitted for participants who initially received capecitabine and oxaliplatin) once every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Oxaliplatin; Drug: Capecitabine; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Tislelizumab — 200 mg intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: BGB-A317; TEVIMBRA®
  Arms: Tislelizumab + Chemotherapy
Drug: Placebo — Placebo to match tislelizumab IV on Day 1 of each 21-day cycle
  Arms: Placebo + Chemotherapy
Drug: Cisplatin — 80 mg/m² IV on Day 1 of each 21-day cycle
Drug: Oxaliplatin — 130 mg/m² IV on Day 1 of each 21-day cycle
Drug: Capecitabine — 1000 mg/m² orally twice daily (BD) Days 1 through 14 (14 days total) of each 21-day cycle
Drug: 5-Fluorouracil — 800 mg/m²/day IV using continuous infusion on Days 1 to 5 of each 21-day cycle

SUMMARY:
This study was designed to compare the efficacy and safety of tislelizumab plus chemotherapy versus placebo plus chemotherapy as the first treatment (first-line) for adults diagnosed with locally advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Locally advanced unresectable or metastatic gastric cancer (GC) or gastroesophageal junction (GEJ) carcinoma and have histologically confirmed adenocarcinoma
2. No previous systemic therapy for locally advanced unresectable or metastatic gastric/GEJ cancer. NOTE: Participants may have received prior neoadjuvant or adjuvant therapy as long as it was completed and have no recurrence or disease progression for at least 6 months.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1 within 7 days prior to randomization
4. Adequate organ function ≤ 7 days prior to randomization

Key Exclusion Criteria:

1. Has squamous cell or undifferentiated or other histological type GC
2. Active leptomeningeal disease or uncontrolled brain metastasis
3. Diagnosed with gastric or GEJ adenocarcinoma with positive HER2
4. Prior therapy with an anti-programmed cell death protein-1 (PD-1), anti-programmed cell death protein ligand-1 (PD-L1), anti-programmed cell death protein ligand-2 (PD-L2), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wang, MD, Study Director — BeiGene
Locations (149):
- United States (6):
  - University of California Davis Health System, Sacramento, California
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Ohio State University Hospital, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
- China (51):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Foshan First Peoples Hospital, Foshan, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Shenzhen Peoples Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital Branch South, Nantong, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (7):
  - Centre Georges Francois Leclerc, Dijon
  - Chu Besancon Hopital Jean Minjoz, Doubs
  - Hopital de La Timone, Marseille
  - Icl Alexis Vautrin, Meurthe Et Moselle
  - Hopital Nord Franche Comte Site Du Mittan, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - Chu Bordeaux Hopital Haut Leveque, Pessac
- Italy (11):
  - Azienda Ospedaliera Universitaria Policlinico Santorsola Malpighi, Bologna
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Nazionale Tumori Fondazione G Pascale, Napoli
  - Iov Istituto Oncologico Veneto Irccs, Padua
  - Ao Ospedali Riuniti Marche Nord, Pesaro
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Irccs Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Aou Senese Policlinico Santa Maria Alle Scotte, Siena
  - Azienda Ospedaliera Citta Della Salute E Della Scienza Di Torino, Torino
  - Azienda Ospedaliera Universitaria Delle Marche, Torrette
- Japan (23):
  - Chiba Cancer Center, Chiba, Chiba
  - Tesshokai Kameda General Hospital, Kamogawashi, Chiba
  - Nho Shikoku Cancer Center, Matsuyama, Ehime
  - Nho Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gunma Prefectural Cancer Center, Otashi, Gunma
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Johas Kansai Rosai Hospital, Amagasakishi, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kitagun, Kagawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Oita University Hospital, Yufushi, Oita Prefecture
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Izumi City General Hospital, Izumishi, Osaka
  - Nho Osaka National Hospital, Osakashi, Osaka
  - Osaka University Hospital, Suitashi, Osaka
  - Saitama Medical University International Medical Center, Hidakashi, Saitama
  - Saitama Cancer Center, Kitaadachigun, Saitama
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsushi, Shizuoka
  - National Cancer Center Hospital, Chuoku, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchushi, Tokyo
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - Center Hospital of the National Center For Global Health and Medicine, Shinjukuku, Tokyo
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Terapii Wspolczesnej Jm Jasnorzewska Sp Komandytowo Akcyjna, Lodz
  - Przychodnia Med Polonia Sp Z Oo, Poznan
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
- Pan American Oncology Trials, Llc, Rio Piedras, Puerto Rico
- Russia (10):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Rbih Ivanovo Regional Oncological Dispensary, Ivanovo, Ivanovo Oblast
  - Vitamed Llc, Moscow, Moscow
  - Sbhi of Novosibirsk Region Novosibirsk Regional Oncological Dispensary, Novosibirsk, Novosibirsk Oblast
  - Bih of Omsk Region Clinical Oncology Dispensary, Omsk, Omsk Oblast
  - Private Educational Institution of Higher Education Medical University Reaviz, Samara, Samaraskaya Oblast'
  - Pavlov First Saint Petersburg State Medical University, SaintPetersburg, Sankt-Peterburg
  - Fsbi Clinical Research and Practical Center For Specialized Medical Care (Oncology), SanktPetersburg, Sankt-Peterburg
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary, Volgograd, Volgograd Oblast
  - Sbih of Yaroslavl Region Regional Clinical Oncological Hospital, Yaroslavl, Yaroslavl Oblast
- South Korea (10):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbukdo
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Chung Ang University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (13):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Universitario de Elche, Elche
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Initia Oncologia, Slp, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Acibadem Adana Hospital, Adana
  - Dr Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Nonu Universitesi Tip Fakultesi, Battalgazi
  - Dicle University Medical Faculty, Diyarbakır
  - Akdeniz University Hospital, Konyaalt
  - Iu C, Clinical Research Excellence Application and Research Center, Stanbul
  - Namik Kemal University, Tekirdağ
  - Karadeniz Tecnical Uni Med Fac, Trabzon
- United Kingdom (2):
  - Velindre Cancer Centre, Cardiff
  - Sarah Cannon Research Institute Uk, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Cruz-Correa M, Oh DY, Kato K, Tabernero J, Bai Y, Shi J, Lee KW, Hirano H, Spigel D, Wyrwicz L, Pazo Cid R, Cubillo Gracian A, Xu Y, Sheng T, Yang S, Xu RH, Moehler M. Tislelizumab + Chemotherapy in Gastric Cancer: Long-Term RATIONALE-305 Randomized Trial Follow-up. Adv Ther. 2026 Jan;43(1):165-183. doi: 10.1007/s12325-025-03415-0. Epub 2025 Nov 18. PMID 41251890
- [Derived] Cruz-Correa M, Xu RH, Moehler M, Oh DY, Kato K, Spigel D, Arkenau HT, Tabernero J, Zimina AV, Bai Y, Shi J, Lee KW, Hirano H, Wyrwicz L, Cid RP, Xu H, Sheng T, Barnes G. Tislelizumab plus chemotherapy versus placebo plus chemotherapy as first-line treatment of advanced gastric or gastroesophageal junction adenocarcinoma: patient-reported outcomes in the RATIONALE-305 study. Curr Med Res Opin. 2025 Jun;41(6):1007-1016. doi: 10.1080/03007995.2025.2501588. Epub 2025 Jun 18. PMID 40528576
- [Derived] Moehler M, Oh DY, Kato K, Arkenau T, Tabernero J, Lee KW, Rha SY, Hirano H, Spigel D, Yamaguchi K, Wyrwicz L, Disel U, Pazo-Cid RA, Fornaro L, Xu Y, Sheng T, Yang S, Kadva A, Cruz-Correa M, Xu RH. First-Line Tislelizumab Plus Chemotherapy for Advanced Gastric Cancer with Programmed Death-Ligand 1 Expression >/= 1%: A Retrospective Analysis of RATIONALE-305. Adv Ther. 2025 May;42(5):2248-2268. doi: 10.1007/s12325-025-03133-7. Epub 2025 Mar 13. PMID 40075025
- [Derived] Li W, Wan L, Zhang J. Cost-effectiveness of tislelizumab plus chemotherapy vs chemotherapy as first-line treatment of PD-L1 positive advanced gastric or gastroesophageal junction adenocarcinoma from a Chinese perspective. Expert Rev Gastroenterol Hepatol. 2024 Jun;18(6):293-301. doi: 10.1080/17474124.2024.2373730. Epub 2024 Jun 28. PMID 38923910
- [Derived] Qiu MZ, Oh DY, Kato K, Arkenau T, Tabernero J, Correa MC, Zimina AV, Bai Y, Shi J, Lee KW, Wang J, Poddubskaya E, Pan H, Rha SY, Zhang R, Hirano H, Spigel D, Yamaguchi K, Chao Y, Wyrwicz L, Disel U, Cid RP, Fornaro L, Evesque L, Wang H, Xu Y, Li J, Sheng T, Yang S, Li L, Moehler M, Xu RH; RATIONALE-305 Investigators. Tislelizumab plus chemotherapy versus placebo plus chemotherapy as first line treatment for advanced gastric or gastro-oesophageal junction adenocarcinoma: RATIONALE-305 randomised, double blind, phase 3 trial. BMJ. 2024 May 28;385:e078876. doi: 10.1136/bmj-2023-078876. PMID 38806195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 141 study centers in 13 countries across Asia, Europe, and North America. Adults with histologically confirmed, locally advanced unresectable or metastatic gastric or gastrooesophageal junction adenocarcinoma and no previous systemic therapy for advanced disease were recruited.
Pre-assignment Details: Participants were randomly assigned to either tislelizumab plus investigator chosen chemotherapy (ICC) or placebo plus ICC.
  Randomization was stratified according to region (China [including Taiwan] vs Japan and South Korea vs Europe/North America), programmed cell death protein ligand-1 (PD-L1) expression (PDL1 tumor area positivity (TAP) score ≥5% or <5%), peritoneal metastases (yes vs no), and investigator's choice of chemotherapy (capecitabine + oxaliplatin, or 5-fluorouracil + cisplatin).
Period: Overall Study
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Started | 501 | 496
Received Treatment | 498 | 494
Completed | 1 | 0
Not Completed | 500 | 496
Not completed — Death | 397 | 431
Not completed — Study Closed by Sponsor | 77 | 38
Not completed — Withdrawal by Subject | 20 | 17
Not completed — Lost to Follow-up | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Tislelizumab + Chemotherapy: Participants received 200 mg of tislelizumab intravenously with investigator's choice of chemotherapy once every 3 weeks for up to six treatment cycles. Thereafter, participants continued treatment with 200 mg tislelizumab, with optional maintenance capecitabine (only permitted for participants who initially received capecitabine and oxaliplatin) once every 3 weeks until disease progression or unacceptable toxicity.
- Placebo + Chemotherapy: Participants received placebo intravenously with investigator's choice of chemotherapy once every 3 weeks for up to six treatment cycles. Thereafter, participants continued treatment with placebo with optional maintenance capecitabine (only permitted for participants who initially received capecitabine and oxaliplatin) once every 3 weeks until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 501 | 496 | 997
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 340 | 313 | 653
  >=65 years | 161 | 183 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.07) | 59.7 (11.20) | 59.3 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 150 | 305
  Male | 346 | 346 | 692
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 492 | 474 | 966
  Unknown or Not Reported | 7 | 16 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 376 | 372 | 748
  White | 116 | 107 | 223
  Not Reported | 8 | 16 | 24
  Other | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Geographic Region [Count of Participants; unit: Participants]
  China (including Taiwan) | 259 | 257 | 516
  Japan and South Korea | 117 | 115 | 232
  North America/Europe | 125 | 124 | 249
Primary Tumor Location [Count of Participants; unit: Participants] — *One participant in the placebo + chemotherapy arm did not report primary location and disease stage, as the diagnosis of this participant was updated from gastric adenocarcinoma to be pancreatic cancer after randomization.
  Participants
    Stomach | 405 | 395 | 800
    Gastro-oesophageal junction | 96 | 100 | 196
    Other* | 0 | 1 | 1
PD-L1 Expression [Count of Participants; unit: Participants] — PDL1 expression was assessed by a central laboratory using the TAP score, defined as total percentage of tumor area (tumor and any desmoplastic stroma) covered by tumor cells with PD-L1 membrane staining (any intensity), and tumor associated immune cells with PD-L1 staining (any intensity), visually estimated by pathologists using an investigational use only version of the Ventana PDL1 (SP263) assay.
  Participants
    < 5% | 227 | 224 | 451
    ≥ 5% | 274 | 272 | 546
Presence of Peritoneal Metastasis [Count of Participants; unit: Participants]
  Yes | 220 | 214 | 434
  No | 281 | 282 | 563
Investigator Chosen Chemotherapy [Count of Participants; unit: Participants]
  Oxaliplatin + Capecitabine | 466 | 465 | 931
  Cisplatin + 5-Fluorouracil | 35 | 31 | 66

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in PD-L1 Positive Participants
Description: Overall survival (OS) is defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up to the primary analysis data cut-off date of 8 October 2021; Median (range) time on follow-up was 11.8 (0.1 - 33.4) months.
Population: The PD-L1-Positive Analysis Set included all randomized participants whose tumors were PD-L1 positive (defined as PD-L1 TAP score ≥ 5%)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 274 | 272
months | 17.2 [13.9 to 21.3] | 12.6 [12.0 to 14.4]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p = 0.0056, One-sided Log Rank Test — The superiority boundary at the primary overall survival analysis was predefined using the O'Brien-Fleming boundary approximated using the Hwang-Shih-DeCani spending function at 0.0092; One-Sided Log-Rank Test stratified by regions (Asia versus Europe/North America) and presence of peritoneal metastasis (yes vs no); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.59 to 0.94] — The stratified hazard ratio and two-sided 95% confidence interval were estimated using a Cox proportional hazard regression model, including treatment arm as a covariate, and region and presence of peritoneal metastasis as strata

2. Primary Outcome: Overall Survival in the Intent-to-Treat (ITT) Analysis Set
Description: as for outcome 1
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 28 February 2023; Median (range) time on follow-up was 13.2 (0.1 - 50.1) months.
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 501 | 496
months | 15.0 [13.6 to 16.5] | 12.9 [12.1 to 14.1]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p = 0.0011, One-Sided Log-Rank Test — The one sided P value boundary for superiority of overall survival in all randomized participants at final analysis was 0.0226 based on 776 actual observed deaths; One-Sided Log-Rank test stratified by region (Asia vs Europe/North America), PD-L1 expression (<5% vs ≥5%), and presence of peritoneal metastasis; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.70 to 0.92] — The stratified hazard ratio and two-sided 95% confidence interval were estimated using a Cox proportional hazard regression model, including treatment arm as a covariate, and region, PD-L1 expression, and presence of peritoneal metastasis as strata

3. Secondary Outcome: Progression-free Survival (PFS) in PD-L1 Positive Participants
Description: Progression-free survival is defined as the time from the date of randomization to the date of the first objectively documented tumor progression assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: PD-L1 Positive Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 274 | 272
months | 7.2 [5.8 to 8.4] | 5.9 [5.6 to 7.0]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.56 to 0.83] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Response Rate (ORR) in PD-L1 Positive Participants
Description: ORR is defined as the percentage of participants whose best overall response is complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors v1.1 assessed by the investigator.
  Investigators conducted assessments of radiological tumor response by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST version 1.1 about every six weeks during the first 48 weeks of the study and every nine weeks thereafter.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Response was assessed every 6 weeks for the first 48 weeks and every 9 weeks thereafter; up to the final efficacy analysis data cut-off date of 28 February 2023; Median (range) time on follow-up was 13.2 (0.1 - 50.1) months.
Population: PD-L1 Positive Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 274 | 272
percentage of participants | 51.5 [45.4 to 57.5] | 42.6 [36.7 to 48.8]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Other; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.04] — Odds ratio between arms weas calculated using the Cochran-Mantel-Haenszel method, stratified by regions (Asia versus Europe/North America) and presence of peritoneal metastasis

5. Secondary Outcome: Progression-free Survival (PFS) in the ITT Analysis Set
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Intent-to-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 501 | 496
months | 6.9 [5.7 to 7.2] | 6.2 [5.6 to 6.9]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.67 to 0.90] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Overall Response Rate (ORR) in the ITT Analysis Set
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 501 | 496
percentage of participants | 47.3 [42.9 to 51.8] | 40.5 [36.2 to 45.0]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Other; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.72] — Odds ratio between arms were calculated using the Cochran-Mantel-Haenszel method, stratified by regions (Asia versus Europe/North America), PD-L1 expression and presence of peritoneal metastasis

7. Secondary Outcome: Duration of Response (DOR) in PD-L1 Positive Participants
Description: DOR is defined as the time from the first determination of an objective response assessed by the investigator per RECIST v1.1, until the first documentation of progression or death, whichever occurred first.
  Progressive disease (PD): At least a 20% increase in the size of target lesions, taking as reference the smallest size on study, with an absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: as for outcome 4
Population: Participants in the PD-L1 Positive Analysis Set with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 141 | 116
months | 10.0 [8.2 to 16.8] | 6.9 [5.7 to 8.5]

8. Secondary Outcome: Duration of Response in the ITT Analysis Set
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Participants in the ITT Analysis Set with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 237 | 201
months | 8.6 [7.9 to 11.1] | 7.2 [6.0 to 8.5]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/Quality of Life (QOL) and Physical Functioning Scores
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed to a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline and Cycles 4 and 6
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-C30 at baseline; participants with available data at baseline and the relevant postbaseline visit are included in the analysis at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 465 | 467
score on a scale
  Global Health Status/QOL: Cycle 4: number analyzed (Participants) | 388 | 380
  Global Health Status/QOL: Cycle 4 | 1.35 [-0.24 to 2.94] | -0.45 [-2.04 to 1.13]
  Global Health Status/QOL: Cycle 6: number analyzed (Participants) | 359 | 339
  Global Health Status/QOL: Cycle 6 | 0.93 [-0.71 to 2.57] | -1.58 [-3.24 to 0.07]
  Physical Functioning: Cycle 4: number analyzed (Participants) | 388 | 380
  Physical Functioning: Cycle 4 | -2.47 [-3.77 to -1.18] | -3.92 [-5.21 to -2.62]
  Physical Functioning: Cycle 6: number analyzed (Participants) | 359 | 339
  Physical Functioning: Cycle 6 | -2.76 [-4.22 to -1.30] | -5.22 [-6.69 to -3.75]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Global Health Status/QoL at Cycle 4; Test type: Other; Least Squares (LS) Mean Difference = 1.80, 95% CI 2-sided [-0.33 to 3.94] — Mixed effect model analysis with QLQ-C30 scores from cycle 1 to 6 as the response variable, and treatment by study visit interaction, baseline mean score and randomization stratification factors as covariates
Statistical Analysis 2: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Global Health Status/QoL at Cycle 6; Test type: Other; LS Mean Difference = 2.52, 95% CI 2-sided [0.29 to 4.74] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Physical Functioning at Cycle 4; Test type: Other; LS Mean Difference = 1.44, 95% CI 2-sided [-0.27 to 3.16]
Statistical Analysis 4: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Physical Functioning at Cycle 6; Test type: Other; LS Mean Difference = 2.46, 95% CI 2-sided [0.49 to 4.43] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Fatigue Score
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed to a 0 to 100 scale via linear transformation. The fatigue symptom scale includes 3 items and ranges from 0 to 100, where higher scores indicate a higher level of symptoms.
Time Frame: Baseline and Cycles 4 and 6
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 465 | 467
score on a scale
  Cycle 4: number analyzed (Participants) | 388 | 380
  Cycle 4 | 1.75 [-0.09 to 3.60] | 3.07 [1.23 to 4.91]
  Cycle 6: number analyzed (Participants) | 359 | 339
  Cycle 6 | 1.71 [-0.32 to 3.75] | 4.73 [2.68 to 6.77]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Fatigue at Cycle 4; Test type: Other; LS Mean Difference = -1.32, 95% CI 2-sided [-3.79 to 1.15] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Fatigue at Cycle 6; Test type: Other; LS Mean Difference = -3.01, 95% CI 2-sided [-5.78 to -0.24] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Gastric Cancer Module QLQ-STO22 (EORTC QLQ-STO22)
Description: EORTC-QLQ-STO22 is a 22-item questionnaire developed to assess QoL of gastric cancer participants. It consists of 5 multi-item subscales: Dysphagia/odynophagia (4 items), Pain/discomfort (3 items), Dietary restrictions (5 items), Upper gastro-intestinal (GI) symptoms (3 items), Specific emotional problems (3 items) and 4 single items. Each question is answered on a scale from 0 (Not at all) to 4 (Very Much), where lower scores indicate fewer symptoms/better QoL.
  Raw scores were transformed to a scale from 0 to 100, where lower scores indicate better QoL.
  The QLQ-STO22 Index score is the mean of the 6 domain scores and 4 single items.
Time Frame: Baseline and Cycles 4 and 6
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-STO22 at baseline; participants with available data at baseline and the relevant postbaseline visit are included in the analysis at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 465 | 467
units on a scale
  Index Score: Cycle 4: number analyzed (Participants) | 387 | 379
  Index Score: Cycle 4 | -1.71 [-2.77 to -0.66] | -0.61 [-1.66 to 0.45]
  Index Score: Cycle 6: number analyzed (Participants) | 358 | 339
  Index Score: Cycle 6 | -1.84 [-2.95 to -0.74] | -0.22 [-1.34 to 0.89]
  Dysphagia/Odynophagia Scale: Cycle 4: number analyzed (Participants) | 387 | 379
  Dysphagia/Odynophagia Scale: Cycle 4 | -2.78 [-3.99 to -1.57] | -1.27 [-2.48 to -0.06]
  Dysphagia/Odynophagia Scale: Cycle 6: number analyzed (Participants) | 358 | 339
  Dysphagia/Odynophagia Scale: Cycle 6 | -2.79 [-3.93 to -1.64] | -2.01 [-3.17 to -0.86]
  Pain/Discomfort Scale: Cycle 4: number analyzed (Participants) | 387 | 379
  Pain/Discomfort Scale: Cycle 4 | -6.88 [-8.39 to -5.36] | -4.64 [-6.16 to -3.13]
  Pain/Discomfort Scale: Cycle 6: number analyzed (Participants) | 358 | 339
  Pain/Discomfort Scale: Cycle 6 | -5.97 [-7.56 to -4.38] | -4.09 [-5.69 to -2.49]
  Dietary Restrictions Scale: Cycle 4: number analyzed (Participants) | 387 | 379
  Dietary Restrictions Scale: Cycle 4 | -0.31 [-1.75 to 1.12] | 0.61 [-0.82 to 2.05]
  Dietary Restrictions Scale: Cycle 6: number analyzed (Participants) | 358 | 339
  Dietary Restrictions Scale: Cycle 6 | -0.25 [-1.79 to 1.30] | 1.08 [-0.48 to 2.63]
  Upper Gastro-Intestinal Symptoms: Cycle 4: number analyzed (Participants) | 387 | 379
  Upper Gastro-Intestinal Symptoms: Cycle 4 | -3.14 [-4.40 to -1.87] | -1.54 [-2.80 to -0.28]
  Upper Gastro-Intestinal Symptoms: Cycle 6: number analyzed (Participants) | 358 | 339
  Upper Gastro-Intestinal Symptoms: Cycle 6 | -3.24 [-4.58 to -1.90] | -1.49 [-2.84 to -0.14]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Index-Score at Cycle 4; Test type: Other; LS Mean Difference = -1.11, 95% CI 2-sided [-2.53 to 0.31] — Mixed effect model analysis with QLQ-STO22 scores from cycle 1 to 6 as the response variable, and treatment by study visit interaction, baseline mean score and randomization stratification factors as covariates
Statistical Analysis 2: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Index-Score at Cycle 6; Test type: Other; LS Mean Difference = -1.62, 95% CI 2-sided [-3.12 to -0.12] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Dysphagia/Odynophagia Scale at Cycle 4; Test type: Other; LS Mean Difference = -1.51, 95% CI 2-sided [-3.13 to 0.11] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Dysphagia/Odynophagia Scale at Cycle 6; Test type: Other; LS Mean Difference = -0.77, 95% CI 2-sided [-2.31 to 0.76] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Pain/Discomfort Scale at Cycle 4; Test type: Other; LS Mean Difference = -2.23, 95% CI 2-sided [-4.26 to -0.20] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Pain/Discomfort Scale at Cycle 6; Test type: Other; LS Mean Difference = -1.88, 95% CI 2-sided [-4.03 to 0.27] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Dietary Restrictions Scale at Cycle 4; Test type: Other; LS Mean Difference = -0.93, 95% CI 2-sided [-2.85 to 0.99] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Dietary Restrictions Scale at Cycle 6; Test type: Other; LS Mean Difference = -1.32, 95% CI 2-sided [-3.42 to 0.77] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Upper Gastro-Intestinal Symptoms at Cycle 4; Test type: Other; LS Mean Difference = -1.59, 95% CI 2-sided [-3.28 to 0.09] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in QLQ-STO22 Upper Gastro-Intestinal Symptoms at Cycle 6; Test type: Other; LS Mean Difference = -1.74, 95% CI 2-sided [-3.55 to 0.06] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in European Quality of Life 5-Dimensions, 5-level (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline and Cycles 4 and 6
Population: Participants in the ITT Analysis Set who completed the EQ-5D-5L at baseline; participants with available data at baseline and the relevant postbaseline visit are included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 465 | 467
score on a scale
  Cycle 4: number analyzed (Participants) | 360 | 364
  Cycle 4 | 2.9 (15.62) | 0.8 (14.91)
  Cycle 6: number analyzed (Participants) | 331 | 322
  Cycle 6 | 3.0 (16.38) | -0.8 (15.17)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drugs, whether related to study drugs or not.
  An SAE is any untoward medical occurrence that, at any dose met any of the following criteria:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the Investigator based on medical judgement.
Time Frame: From first dose of study drug to 30 days after last dose or the initiation of a new anticancer therapy, whichever occurred first, up to the end of study; maximum treatment duration was 59.3 months in Tislelizumab and 56.8 months in the Placebo group.
Population: The Safety Analysis Set included all participants who received ≥ 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 498 | 494
Participants
  Any TEAE | 495 | 486
  Any SAE | 211 | 179

14. Secondary Outcome: Disease Control Rate in PD-L1 Positive Participants
Description: Disease Control Rate is defined as the percentage of participants who had confirmed CR, PR, or stable disease (SD) assessed by the investigator and the investigator per RECIST v1.1. Investigators conducted assessments of radiological tumor response by CT or MRI per RECIST version 1.1 about every six weeks during the first 48 weeks of the study and every nine weeks thereafter.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
  SD: Neither sufficient shrinkage in size of lesions to qualify for PR nor sufficient increase to qualify for PD, and no new lesions.
Time Frame: as for outcome 4
Population: PD-L1 Positive Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 274 | 272
percentage of participants | 88.3 [83.9 to 91.9] | 83.1 [78.1 to 87.3]

15. Secondary Outcome: Disease Control Rate in the ITT Analysis Set
Description: Disease Control Rate is defined as the percentage of participants who had confirmed CR, PR, or stable disease (SD) assessed by the investigator per RECIST v1.1. Investigators conducted assessments of radiological tumor response by CT or MRI per RECIST version 1.1 about every six weeks during the first 48 weeks of the study and every nine weeks thereafter.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
  SD: Neither sufficient shrinkage in size of lesions to qualify for PR nor sufficient increase to qualify for PD, and no new lesions.
Time Frame: as for outcome 4
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 501 | 496
percentage of participants | 89.8 [86.8 to 92.3] | 83.3 [79.7 to 86.4]

16. Secondary Outcome: Clinical Benefit Rate (CBR) in PD-L1 Positive Participants
Description: Clinical benefit rate is defined as the percentage of participants who achieved a confirmed complete response, partial response, or durable stable disease assessed by the Investigator per RECIST v1.1.
  CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, persistence of one or more nontarget lesion(s) and/or maintenance of tumor marker level above the normal limits.
  Durable SD: Stable disease for ≥ 24 weeks.
Time Frame: as for outcome 4
Population: PD-L1 Positive Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 274 | 272
percentage of participants | 65.0 [59.0 to 70.6] | 59.2 [53.1 to 65.1]

17. Secondary Outcome: Clinical Benefit Rate (CBR) in the ITT Analysis Set
Description: as for outcome 16
Time Frame: as for outcome 4
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 501 | 496
percentage of participants | 63.1 [58.7 to 67.3] | 58.9 [54.4 to 63.2]

18. Secondary Outcome: Time to Response (TTR) in PD-L1 Positive Participants
Description: Time to response is defined as the time from randomization to the first determination of an objective response per RECIST version 1.1 as assessed by the investigator.
Time Frame: as for outcome 2
Population: Participants in the PD-L1 Positive Analysis Set with an objective response
Measure: Median (Full Range); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 141 | 116
months | 1.4 [0.9 to 11.3] | 1.4 [1.0 to 17.5]

19. Secondary Outcome: Time to Response (TTR) in the ITT Analysis Set
Description: as for outcome 18
Time Frame: as for outcome 2
Population: Participants in the ITT Analysis Set with an objective response
Measure: Median (Full Range); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 237 | 201
months | 1.4 [0.9 to 13.4] | 1.4 [1.0 to 17.5]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose or the initiation of a new anticancer therapy, whichever occurred first, up to the end of study; maximum treatment duration was 59.3 months in Tislelizumab and 56.8 months in the Placebo group.
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 397/501 | 431/496
Serious Adverse Events (participants affected / at risk) | 211/498 | 179/494
Other Adverse Events (participants affected / at risk) | 489/498 | 485/494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Chemotherapy (N=498) | Placebo + Chemotherapy (N=494)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 10 (10)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (5)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 5 (5) | 5 (5)
Bezoar (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 3 (4)
Gastric haemorrhage (Gastrointestinal disorders) | 6 (7) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 5 (5) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ischaemic enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 5 (6)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 7 (8)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 5 (5)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 10 (10) | 5 (5)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 1 (1)
General physical health deterioration (General disorders) | 6 (6) | 7 (7)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Polyserositis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 6 (6)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 6 (7) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 5 (5) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 4 (4)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Immune-mediated adverse reaction (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (3) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 12 (13) | 14 (18)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Remnant gastritis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Fibrin degradation products increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 16 (21) | 17 (21)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint adhesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary tumour thrombotic microangiopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 4 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Immune-mediated renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Chemotherapy (N=498) | Placebo + Chemotherapy (N=494)
Anaemia (Blood and lymphatic system disorders) | 197 (374) | 202 (355)
Leukopenia (Blood and lymphatic system disorders) | 44 (193) | 45 (123)
Neutropenia (Blood and lymphatic system disorders) | 75 (247) | 82 (184)
Thrombocytopenia (Blood and lymphatic system disorders) | 64 (131) | 56 (101)
Hypothyroidism (Endocrine disorders) | 63 (73) | 13 (13)
Cataract (Eye disorders) | 18 (21) | 22 (25)
Abdominal discomfort (Gastrointestinal disorders) | 16 (23) | 8 (9)
Abdominal distension (Gastrointestinal disorders) | 53 (61) | 52 (59)
Abdominal pain (Gastrointestinal disorders) | 75 (109) | 80 (97)
Abdominal pain upper (Gastrointestinal disorders) | 51 (62) | 55 (80)
Ascites (Gastrointestinal disorders) | 18 (18) | 9 (10)
Constipation (Gastrointestinal disorders) | 90 (123) | 105 (144)
Diarrhoea (Gastrointestinal disorders) | 134 (223) | 144 (241)
Dry mouth (Gastrointestinal disorders) | 23 (28) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 21 (21) | 28 (37)
Dysphagia (Gastrointestinal disorders) | 21 (23) | 17 (20)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 (20) | 26 (38)
Nausea (Gastrointestinal disorders) | 248 (469) | 237 (443)
Stomatitis (Gastrointestinal disorders) | 37 (47) | 35 (44)
Vomiting (Gastrointestinal disorders) | 176 (330) | 178 (352)
Asthenia (General disorders) | 97 (121) | 86 (116)
Chest discomfort (General disorders) | 15 (17) | 11 (18)
Chills (General disorders) | 20 (26) | 7 (7)
Fatigue (General disorders) | 87 (105) | 73 (101)
Malaise (General disorders) | 37 (45) | 41 (49)
Oedema peripheral (General disorders) | 41 (48) | 38 (42)
Pyrexia (General disorders) | 99 (185) | 66 (92)
COVID-19 (Infections and infestations) | 20 (27) | 14 (14)
Pneumonia (Infections and infestations) | 19 (19) | 13 (14)
Upper respiratory tract infection (Infections and infestations) | 25 (34) | 13 (15)
Alanine aminotransferase increased (Investigations) | 123 (188) | 105 (175)
Aspartate aminotransferase increased (Investigations) | 157 (285) | 150 (274)
Blood alkaline phosphatase increased (Investigations) | 19 (33) | 22 (25)
Blood bilirubin increased (Investigations) | 75 (171) | 74 (172)
Blood creatine phosphokinase increased (Investigations) | 17 (30) | 20 (32)
Blood creatinine increased (Investigations) | 15 (22) | 14 (16)
Blood lactate dehydrogenase increased (Investigations) | 18 (36) | 20 (33)
Gamma-glutamyltransferase increased (Investigations) | 19 (31) | 22 (27)
Lymphocyte count decreased (Investigations) | 28 (67) | 22 (45)
Neutrophil count decreased (Investigations) | 172 (705) | 163 (573)
Platelet count decreased (Investigations) | 173 (384) | 184 (390)
Weight decreased (Investigations) | 110 (139) | 102 (122)
Weight increased (Investigations) | 28 (36) | 9 (9)
White blood cell count decreased (Investigations) | 120 (580) | 136 (488)
Decreased appetite (Metabolism and nutrition disorders) | 202 (277) | 207 (327)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (17) | 15 (23)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 87 (147) | 92 (130)
Hypocalcaemia (Metabolism and nutrition disorders) | 22 (24) | 11 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 84 (152) | 57 (89)
Hyponatraemia (Metabolism and nutrition disorders) | 36 (54) | 31 (38)
Hypoproteinaemia (Metabolism and nutrition disorders) | 21 (25) | 25 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 24 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (35) | 40 (46)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 18 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (22) | 22 (23)
Dizziness (Nervous system disorders) | 41 (54) | 42 (52)
Dysgeusia (Nervous system disorders) | 25 (29) | 18 (18)
Headache (Nervous system disorders) | 20 (23) | 19 (21)
Hypoaesthesia (Nervous system disorders) | 70 (99) | 69 (110)
Neurotoxicity (Nervous system disorders) | 13 (23) | 16 (27)
Paraesthesia (Nervous system disorders) | 12 (12) | 18 (25)
Peripheral sensory neuropathy (Nervous system disorders) | 106 (134) | 118 (156)
Insomnia (Psychiatric disorders) | 47 (51) | 53 (65)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (34) | 32 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (37) | 33 (41)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 16 (23)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 20 (24)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 95 (107) | 93 (111)
Pruritus (Skin and subcutaneous tissue disorders) | 52 (65) | 15 (19)
Rash (Skin and subcutaneous tissue disorders) | 43 (52) | 17 (19)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 20 (21) | 14 (16)
Hypertension (Vascular disorders) | 12 (21) | 23 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03777657/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03777657/SAP_001.pdf